CLINICAL TRIAL: NCT06984549
Title: Telemedicine for Evaluating Dry Eye Disease (DED) Using a Mobile Phone-Attached Portable Automatic Ocular Surface Imaging Device (PAOSID): A Patient-Operated Diagnostic and Continuous Ocular Surface Monitoring (COSM) System
Brief Title: Telemedicine Evaluation of Dry Eye Disease Using a Portable Automatic Ocular Surface Imaging Device (PAOSID)
Status: Recruiting | Type: Observational
Sponsor: Chen Wei (Other)
Collaborators: Singapore National Eye Centre (Other Government); University of Sydney (Other)
Responsible Party: Sponsor-Investigator, Chen Wei, Sponsor-Investigator, The Eye Hospital of Wenzhou Medical University
Organization: The Eye Hospital of Wenzhou Medical University (Other)
Other Study IDs: ChiCTR2500097802; 263551 (Registry Identifier: Chinese Clinical Trial Registry (ChiCTR))
Record Dates: First submitted 2025-05-11; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- DED group
  Interventions: Other: DED diagnosis using PAOSID; Other: DED diagnosis using slit lamp
- healthy control
  Interventions: Other: DED diagnosis using PAOSID; Other: DED diagnosis using slit lamp

INTERVENTIONS:
Other: DED diagnosis using PAOSID — A non-invasive diagnostic approach using the Portable Automatic Ocular Surface Imaging Device (PAOSID) to capture anterior segment images and videos for the assessment of dry eye disease (DED).
Other: DED diagnosis using slit lamp — A non-invasive diagnostic approach using the slit lamp to capture anterior segment images and videos for the assessment of dry eye disease (DED).

SUMMARY:
This study aims to evaluate the diagnostic accuracy and grading consistency of a mobile phone-attached portable automatic ocular surface imaging device (PAOSID) for assessing dry eye disease (DED). Both patients diagnosed with DED and healthy volunteers will undergo conventional clinical imaging, including white-light anterior segment photography, corneal fluorescein staining (CFS) under cobalt blue light, and tear film break-up time (TBUT), all performed under slit-lamp examination, as well as meibography. Clinical grading of DED severity will follow the TFOS DEWS I criteria, while other ocular surface findings-such as conjunctival injection, meibomian gland area loss, and CFS-will be assessed using standard ocular surface disease scoring scales.

Following the clinical assessment, participants will use the PAOSID device to independently capture similar ocular surface images and videos. These remote images and videos will first be used to determine whether the participant has dry eye disease (DED). Regardless of the diagnosis result, all participants will undergo severity grading based on the TFOS DEWS I criteria, along with standardized scoring of ocular surface conditions such as conjunctival injection, meibomian gland area loss, and corneal fluorescein staining (CFS). The study will compare remote and clinical assessments to evaluate diagnostic agreement and grading consistency, and assess patient satisfaction and usability of the PAOSID system.

DETAILED DESCRIPTION:
Multicenter, Cross-sectional

ELIGIBILITY:
Inclusion Criteria:

1. Participants included individuals with dry eye, based on the TFOS DEWS II (The Tear Film and Ocular Surface Society Dry Eye Workshop II) guidelines,(19) as well as relatively healthy individuals with no ocular conditions who voluntarily agreed to participate in the study.
2. Participants, or their companions or caregivers, who are willing and able to use the study smartphone to capture relevant eye images and videos.
3. Aged 18 years or older.
4. Provide informed consent.

Exclusion Criteria:

1. Participants with ocular surface disorders other than DED that may affect the appearance of the ocular surface (e.g., pterygium, keratitis, corneal scarring) or with any organic pathologies impacting vision (e.g., cataracts, glaucoma, retinal diseases).
2. Patients currently wearing scleral lenses or bandage contact lenses.
3. Unable to cooperate with the PAOSID, such as due to a serious mental illness or brain damage causing loss of limb control.
4. Significant changes in the ocular images since diagnosis due to factors such as postdiagnostic treatment.

Eye selection criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes patients clinically diagnosed with dry eye disease (DED) and age-matched healthy volunteers. All participants undergo both PAOSID-based and slit-lamp-based ocular surface imaging for diagnostic and grading comparison.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between PAOSID-based and slit-lamp-based DED diagnosis | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- The Eye Hospital, Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided